CLINICAL TRIAL: NCT04879472
Title: Early Functional Outcome of Operative Treatment of Displaced Femoral Neck Fractures in Two Kenyan Orthopaedic Centres
Status: Completed | Type: Observational
Sponsor: University of Nairobi (Other)
Responsible Party: Principal Investigator, Sephenia Raduma Ochieng, Principal Investigator, University of Nairobi
Other Study IDs: UniNairobi
Record Dates: First submitted 2021-05-01; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Fracture Neck of Femur; Hip Fracture; Femoral Neck Fracture
Keywords: Hip fracture; Fracture neck femur; Osteosynthesis; Arthroplasty; Functional outcome
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures | interventions — Fracture Fixation, Internal; Hemiarthroplasty; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Age 50 years and below: 1. Type of surgery (modality of treatment) either osteosynthesis, Hemiarthroplasty or Total hip replacement
  2. Surgical approach either posterior, lateral or anterolateral
  3. Type of anaesthesia either general or spinal
  4. Presence or absence of comorbidities
  5. Sex
  Interventions: Procedure: Osteosynthesis
- Age more than 50 years: 1. Type of surgery (modality of treatment) either osteosynthesis, Hemiarthroplasty or Total hip replacement
  2. Surgical approach either posterior, lateral or anterolateral
  3. Type of anaesthesia either general or spinal
  4. Presence or absence of comorbidities
  5. Sex
  Interventions: Procedure: Osteosynthesis

INTERVENTIONS:
Procedure: Osteosynthesis — The elderly are mainly treated by arthroplasty (total hip replacement or hemiarthroplasty) while the younger age groups, by osteosynthesis either using pins, screws or nails
  Other Names: Hemiarthroplasty; Total hip replacement

SUMMARY:
This was a prospective cohort study. The study was conducted in the two hospitals after approval by the KNH/UON ethical committee and the board of management of Kikuyu Mission Hospital. Trained data clerks were used for retrieval of data from the respective hospitals with follow-up conducted in the respective clinics and through phone calls. The clerks were not blinded to the study but every data was corroborated by interviewing the patients or their relatives and evaluation of medical data availed as well as clinical status. Both KNH and Kikuyu Mission Hospitals had handwritten patient notes/records at the time of the study (not electronic) with central registries for storage of patient files. The patients files and other medical documents will be available in the wards but upon discharge, stored at the central registries.

The WOMAC scores(assessment of the outcome measures) were conducted by the principal investigator by direct interview of the patients/ their designated next of kin, or via telephone contacts. The outcome measures included pain, stiffness and activities of daily living.

DETAILED DESCRIPTION:
This was a prospective cohort study.

The study was conducted in the two hospitals after approval by the Kenyatta National Hospital (KNH)/University of Nairobi (UON) ethical committee and the board of management of Kikuyu Mission Hospital (KMH). Trained data clerks were used for retrieval of data from the respective hospitals with follow-up conducted in the respective clinics and through phone calls. The clerks were not blinded to the study but every data was corroborated by interviewing the patients or their relatives and evaluation of medical data availed as well as clinical status. Both KNH and Kikuyu Mission Hospitals had handwritten patient notes/records at the time of the study (not electronic). Both institutions respectively maintained central registries for storage of patient files following discharge from inpatient care. At the time of the study, this were a hybrid of electronic and manual data storage systems as the electronic system was being introduced. The patients files and other medical documents will be available in the wards but upon discharge, stored at the central registries.

The Western Ontario and MacMaster Universities Osteoarthritis Index (WOMAC) scores were conducted by the principal investigator by direct interview of the patients/ their designated next of kin, or via telephone contacts. This was for the assessment of the outcome measures that included pain, stiffness and activities of daily living. The measures were accessed for the period within two weeks before injury, for the pre-injury functional status and at three months after injury for the early functional status.

This study has been completed and results available.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age and above who underwent operative treatment of displaced fracture neck of femur in the two institutions during the study period.
* Written informed consent.

Exclusion Criteria:

* Patients who had un-displaced or bilateral fracture neck of femur, concomitant pelvic or lower limb fracture/ dislocation, multiple injuries, confusion, previous ipsilateral FNF or FNF surgery, operative treatment done outside the study setting, malignant/ pathological fractures or peri-prosthetic fractures;
* Patients who were non-ambulatory prior to injury and those with chronic pain syndrome and/ or chronic opioid use;
* Patients who declined to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included those patients 18 years of age and above who underwent operative treatment of displaced fracture neck of femur at either Kenyatta National Hospital or Kikuyu Mission Hospital during the study period with granted written informed consent; except those with un-displaced or bilateral fracture neck of femur, concomitant pelvic or lower limb fracture/ dislocation, multiple injuries, confusion, previous ipsilateral FNF or FNF surgery, operative treatment done outside the study setting, malignant/ pathological fractures or peri-prosthetic fractures; those non-ambulatory prior to injury and those with chronic pain syndrome and/ or chronic opioid use.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-11-12 (Actual); Primary Completion 2009-05-11 (Actual); Study Completion 2009-05-11 (Actual)

PRIMARY OUTCOMES:
Pain score | within two weeks of assessment
  Pre-injury pain score in Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index compared with three months' post-operative pain score. The scores are normalised into a scale of 0-100 with 100 indicating no pain and 0, worst pain disability.
Stiffness score | within two weeks of assessment
  Pre-injury Stiffness score in Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index compared with three months' post-operative Stiffness score. The scores are normalised into a scale of 0-100 with 100 indicating no Stiffness disability and 0, worst stiffness disability
Activities of daily living (ADL) score | within two weeks of assessment
  Pre-injury Activities of Daily living(ADL) score in Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index compared with three months' post-operative Activities of Daily living(ADL) score. The scores are normalised into a scale of 0-100 with 100 indicating best Activities of Daily living(ADL) and 0, poor performance in Activities of Daily living(ADL)

SECONDARY OUTCOMES:
Length of hospital stay | three months
  duration of inpatient care

CONTACTS AND LOCATIONS:
Overall Officials: SEPHENIA R OCHIENG', MBChB, MMed, MCh., Principal Investigator — University of Nairobi; JOHN E O ATING'A, MBChB, MCh, Study Director — University of Nairobi; KIRSTINGS A ONDIKO, MBChB, MMed, FCS, Study Director — University of Nairobi; JOHN KINGORI, MBChB, MMed, Study Director — University of Nairobi/ Kikuyu Mission Hospital

IPD SHARING:
Plan to Share IPD: Yes
Share the study protocol, methodology and findings with other researches
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: six years, renewable
Access Criteria: email contact to the principal investigator

REFERENCES:
- [Result] Ochieng SR, Kingori J, Awori KO, Ating'a JEO. Recovery of pre-injury functional state following operative treatment of displaced femoral neck fractures; a prospective cohort study. Ann Med Surg (Lond). 2021 Aug 11;69:102682. doi: 10.1016/j.amsu.2021.102682. eCollection 2021 Sep. PMID 34429951

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2009-05-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT04879472/Prot_SAP_ICF_000.pdf